CLINICAL TRIAL: NCT01106196
Title: The Role of Influenza as a Trigger for Acute Myocardial Infarction: a Self-controlled Case Series Analysis of Linked Data From the Myocardial Ischaemia National Audit Project (MINAP) and the General Practice Research Database (GPRD)
Brief Title: The Role of Influenza as a Trigger for Acute Myocardial Infarction: a CALIBER Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Open University (Other)
Responsible Party: Principal Investigator, Charlotte Warren-Gash, Dr, University College, London
Other Study IDs: CALIBER 09-08; Ref G0800689, no. 87420 (Other Grant/Funding Number: Medical Research Council); Ref 086091/Z/08/Z (Other Grant/Funding Number: Wellcome grant)
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Myocardial Infarction; Influenza
Keywords: Influenza, Human; Influenza, Human/complications; Myocardial infarction/etiology; Cardiovascular Diseases/mortality
MeSH Terms: conditions — Myocardial Infarction; Influenza, Human; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MI plus respiratory illness: Patients with an incident myocardial infarction who also have a record of a visit to primary care with a respiratory tract infection

SUMMARY:
The purpose of this study is to examine the incidence of acute myocardial infarction (MI) occurring after an influenza-like illness using linked primary care and disease registry databases.

DETAILED DESCRIPTION:
This study will measure the incidence ratio for MI occurring in time periods after presentation with an acute respiratory illness compared to baseline time periods using the self-controlled case series method, with reference to the timing of the influenza season (defined by national virological and clinical surveillance data). It will also validate accuracy and completeness of information on MI in the GPRD using linked anonymised data from both MINAP and Hospital Episode Statistics.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be registered with a GPRD 'up to standard' practice during the study period 01/01/1999-31/12/2008
* They must have a record of an incident myocardial infarction (defined by a Read codelist submitted to and agreed by GPRD) that occurs both within their registration and the study period
* They must have at least 6 months between their registration date and the date of the incident MI
* They must have accessed primary care on at least one occasion for a respiratory illness during the study period

Exclusion Criteria:

* Not fulfilling above criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an incident myocardial infarction who also have a record of a visit to primary care with a respiratory tract infection occurring within the study period (01/01/99 - 31/12/2008)
Sampling Method: Non-Probability Sample
Enrollment: 11208 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence ratio for acute MI | 28 days
  Incidence ratio for MI occurring in time periods after presentation to primary care with an acute respiratory illness compared to baseline time periods

CONTACTS AND LOCATIONS:
Overall Officials: Harry Hemingway, FRCP, Study Director — UCL
Locations (2):
- United Kingdom (2):
  - University College London (UCL), London, London
  - London School of Hygiene & Tropical Medicine, London, London

REFERENCES:
- [Derived] Warren-Gash C, Hayward AC, Hemingway H, Denaxas S, Thomas SL, Timmis AD, Whitaker H, Smeeth L. Influenza infection and risk of acute myocardial infarction in England and Wales: a CALIBER self-controlled case series study. J Infect Dis. 2012 Dec 1;206(11):1652-9. doi: 10.1093/infdis/jis597. Epub 2012 Oct 9. PMID 23048170